CLINICAL TRIAL: NCT03628599
Title: Two Daily Disposable Contact Lenses in Symptomatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLS312-P001
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Myopia
Keywords: Symptomatic
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TOTAL1 (Experimental): Delefilcon A contact lenses worn bilaterally (in both eyes) for 4 weeks in a daily disposable modality
  Interventions: Device: Delefilcon A contact lenses
- 1-DAY (Active Comparator): Senofilcon A contact lenses worn bilaterally for 4 weeks in a daily disposable modality
  Interventions: Device: Senofilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Water Gradient silicon hydrogel daily disposable contact lenses
  Other Names: DAILIES TOTAL1® (DT1)
  Arms: TOTAL1
Device: Senofilcon A contact lenses — Silicon hydrogel daily disposable contact lenses with HydraLuxe™ Technology
  Other Names: ACUVUE OASYS® 1-DAY
  Arms: 1-DAY

SUMMARY:
The purpose of this study is to evaluate the performance of DAILIES TOTAL1® and ACUVUE OASYS® 1-DAY and with respect to visual acuity in a symptomatic study population of monthly or bi-weekly replacement lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and must sign an IRB-approved informed consent form;
* Soft contact lens wearers in both eyes during the past 3 months;
* Best-corrected visual acuity (BCVA) 20/25 or better in each eye;
* Willing to wear study lenses at least 3 days per week and at least 8 hours per day;
* Willing to stop wearing habitual contact lenses for the duration of study participation.

Exclusion Criteria:

* Infection, inflammation, abnormality, condition, disease, surgery, or use of medications, as specified in the protocol;
* Intolerance, hypersensitivity, or allergy to any component of the study products;
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Monocular (only one eye with functional vision).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (4):
- United States (4):
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Pittsburg, Kansas
  - Alcon Investigative Site, Powell, Ohio
  - Alcon Investigative Site, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 investigational sites located in the United States.
Pre-assignment Details: Of the 39 enrolled, 2 subjects were discontinued (1 screen failure, 1 due to lens power not available) prior to randomization. This reporting group includes all randomized subjects (37).
Period: Overall Study
Arm/Group | TOTAL1 | 1-DAY
Started | 18 | 19
Completed | 18 | 18
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any test or control product evaluated in the study (Safety Analysis Set).
Groups:
- TOTAL1: Delefilcon A contact lenses worn bilaterally for 4 weeks in a daily disposable modality
- Total: Total of all reporting groups
Arm/Group | TOTAL1 | 1-DAY | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.4) | 36.9 (9.2) | 36.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 6 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 18 | 36
  Black or African American | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular Corrected Distance Visual Acuity (VA)
Description: Monocular (each eye) corrected (with spectacles or other visual corrective devices) VA was performed under dimmed room illumination using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart at distance. VA was reported in logMAR ("logarithm of the minimum angle of resolution"), with a lower logMAR indicating better visual acuity. No inferential hypotheses was planned for this endpoint.
Time Frame: Week 4
Population: Safety Analysis Set with non-missing response
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | TOTAL1 | 1-DAY
Number analyzed (Participants) | 18 | 18
Number analyzed (Eyes) | 36 | 36
logMAR | -0.01 (0.04) | -0.02 (0.05)

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 4 weeks
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the study lenses. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Safety Analysis Set. "At Risk" population for ocular AEs is included with unit of "eyes."
Groups:
- TOTAL1 Ocular - Right Eye: Right eyes exposed to delefilcon A contact lenses
- TOTAL1 Ocular - Left Eye: Left eyes exposed to delefilcon A contact lenses
- TOTAL1 Non-ocular: All subjects exposed to delefilcon A contact lenses
- 1-DAY Ocular - Right Eye: Right eyes exposed to senofilcon A contact lenses
- 1-DAY Ocular - Left Eye: Left eyes exposed to senofilcon A contact lenses
- 1-DAY Non-ocular: All subjects exposed to senofilcon A contact lenses
Arm/Group | TOTAL1 Ocular - Right Eye | TOTAL1 Ocular - Left Eye | TOTAL1 Non-ocular | 1-DAY Ocular - Right Eye | 1-DAY Ocular - Left Eye | 1-DAY Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 1/19 | 1/19 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL1 Ocular - Right Eye (N=18) | TOTAL1 Ocular - Left Eye (N=18) | TOTAL1 Non-ocular (N=18) | 1-DAY Ocular - Right Eye (N=19) | 1-DAY Ocular - Left Eye (N=19) | 1-DAY Non-ocular (N=19)
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival disorder (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03628599/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT03628599/SAP_001.pdf